CLINICAL TRIAL: NCT06184152
Title: Contrast Ultrasound vs. Abbreviated MRI for Detection of HCC in Patients With Indeterminate Liver Nodules
Brief Title: CEUS vs. AMRI for HCC Detection in Patients With Indeterminate Liver Nodules
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Amit Singal, Lead Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1U01CA283935 (NIH)
Record Dates: First submitted 2023-12-04; First posted 2023-12-28 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-04

CONDITIONS: HCC; Hepatocellular Carcinoma
Keywords: LR3; LR4; HCC Surveillance
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Masking Description: Intervention is not masked for study team or investigator but all images are being interpreted by radiologist who is masked to clinical outcomes (development of HCC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ILN Cohort (Other): Patients with LR3 observations would undergo CEUS and AMRI every 6 months; patients with LR4 observations would undergo CEUS and AMRI 3 months after enrollment and every 6 months thereafter. CEUS and AMRI will preferably be done the same day to minimize burden on the patient, although will be permitted to be completed within 14 days of each other. This interval is sufficiently short to minimize the chance of intervening events. AMRI and CEUS will be performed every 3-6 months until HCC development, regression to LR-1 or LR-2 (i.e., definitely or likely benign, respectively), or end of follow-up at 24 months post-enrollment.
  Interventions: Diagnostic Test: CEUS imaging; Diagnostic Test: aMRI imaging

INTERVENTIONS:
Diagnostic Test: CEUS imaging — Contrast-enhanced ultrasound (CEUS)
Diagnostic Test: aMRI imaging — contrast enhanced abbreviated MRI (AMRI)

SUMMARY:
The study will be conducted at the following locations:

1. UT Southwestern Medical Center
2. Parkland Health and Hospital System
3. University of Michigan

Investigators will prospectively compare the performance of dynamic contrast enhanced abbreviated MRI (AMRI) and contrast-enhanced ultrasound for early-stage HCC detection in patients with indeterminate liver nodules.

DETAILED DESCRIPTION:
Investigators will prospectively perform both abbreviated MRI and contrast-enhanced ultrasound in enrolled patients every 3-6 months. Contrast-enhanced ultrasound and abbreviated MRI will preferably be done the same day, although will be permitted to be completed within 30 days of each other. Abbreviated MRI and contrast-enhanced ultrasound will be performed every 3-6 months until HCC development, regression to LR-1 or LR-2 (i.e., definitely or likely benign, respectively), or end of follow-up at 24 months post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Child A or B cirrhosis from any etiology with at least one ILN on 4-phase CT, contrast- enhanced MRI, or contrast enhanced US but without HCC at baseline.
* Adults 18 years old and above

Exclusion Criteria:

* Patients post liver transplantation
* Patients with concurrent or prior HCC (LR-5 or biopsy proven)
* other liver cancer including cholangiocarcinoma
* Patients with any active extra-hepatic malignancy
* Patients with significant comorbidity and limited life expectancy, e.g., stage D congestive heart failure, in whom surveillance is not warranted are also excluded given unlikely clinical benefit
* Patients with contraindication to contrast-enhanced MRI or CEUS, including implanted medical devices that are considered MR unsafe and severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2028-11-28 (Estimated); Study Completion 2028-11-28 (Estimated)

PRIMARY OUTCOMES:
Early HCC Detection | 5 years
  Assess and compare true positive rate (TPR) and false positive rate (FPR) of AMRI to CEUS for early-stage HCC detection, as defined by the Barcelona Clinic Liver Staging system.

SECONDARY OUTCOMES:
HCC Detection | 5 years
  Evaluate TPR and FPR for any-stage HCC.
Early HCC Detection | 5 years
  Assess and compare true positive rate (TPR) and false positive rate (FPR) of AMRI to CEUS for early-stage HCC detection, as defined by the Milan Criteria

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - University of Texas Southwestern Medical Center, Dallas, Texas